CLINICAL TRIAL: NCT04493034
Title: A Randomized Controlled Trial to Assess the Benefit of Art & Music Therapy on Quality of Life in Patients With Breast Cancer
Brief Title: Assessing the Benefit of Art & Music Therapy on Quality of Life in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5120
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer
Keywords: Cancer Survivors; Music Therapy; Art Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Art Therapy; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Art Therapy (Experimental): Weekly sessions, alternating: in-person sessions (6 over 3 months), home assignments (6 over 3 months)
  Interventions: Behavioral: Art Therapy
- Music Therapy (Experimental): Weekly sessions, alternating: in-person sessions (6 over 3 months), home assignments (6 over 3 months)
  Interventions: Behavioral: Music Therapy
- Standard Of Care (No Intervention): A list of support services is provided. No requirement to attend sessions and no home assignments

INTERVENTIONS:
Behavioral: Art Therapy — The art therapist will assist each participant in producing a bound collection of participant art works/writings for personal, group and/or caregiver inspiration, at the participant's request. For in-person sessions, a variety of studio-based art and writing materials will be available for participant selection and creation. Each session will be directed in the following manner:
  * New therapeutic prompt or bridge from prior session
  * Creative expression, opportunity for reflection, verbal sharing / processing, and a session summary
  * Discussion of action plan for the next consecutive, at-home session (weekly assignment).
  Possible wellness themes for each session (in-person or at-home) may include: mental health, physical health, emotional health, spiritual health, relational health (family and social), or occupational health/financial health.
  Arms: Art Therapy
Behavioral: Music Therapy — Participants have the opportunity to engage in: learning an instrument, active music-making, receptive music-listening, singing, improvisation, song-writing, education on music technology, or music discussion. During in-person musical sessions the six psychosocial goals promoted by the music therapist include: 1) self-care/self-love, 2) support systems, 3) practicing positivity 4) gratitude 5) mindfulness/living in the moment, and 6) goal-setting.
  For at-home assignments, participants will be asked to pick a song of the week that coincides with the theme/goal discussed in previous session(s). They will be asked to write a journal entry about the topic discussed. Journal entries can be freely written or a prompt/question can be provided. If participants do not have access to search for songs or listen to music as at home, they may select a piece from the session and be given lyrics and/or a recording on an .mp3 player returned at conclusion of study.
  Arms: Music Therapy

SUMMARY:
This is a study of art-based and music-based therapy programs lasting three months (with additional follow-up 3 months after the end of the trial) in breast cancer patients currently receiving therapy as well as in cancer survivors.

DETAILED DESCRIPTION:
A cancer diagnosis is often associated with adverse psychosocial effects, including: increased stress and anxiety, fatigue and sleep disturbance, impaired memory and cognition, and poor quality of life. Chemotherapy can cause a cognitive decline in up to 75% of patients; an impairment that oftentimes persists beyond completion of the regimen. This is known as "chemobrain". Integrative therapies are actively being investigated to help improve psychological wellbeing among cancer patients and survivors.

The current standard at this institution is to inform patients of different complementary services that are available, including art therapy, music therapy or acupuncture, but not require patients to use them.

Participants in this study will be randomized to one of three arms 1) Art therapy program, 2) Music therapy program, or 3) Standard of care (SOC). In-person and at-home therapy sessions will be scheduled in alternating, weekly sessions, to allow one week of self-reflection and remote therapy between in-person sessions. Each participant will be asked to attend two in-person therapy sessions per month (total of 6).

The primary objective of this study is to determine the efficacy of a 3-month, therapist-led art or music therapy program to improve quality of life in breast cancer patients currently receiving therapy and in cancer survivors.

Secondary objectives of this study are:

To determine the effect of these programs on patient cognition in this population.

To determine the effect of these programs symptoms of anxiety and depression in this population.

To assess whether the effect of these programs is sustained at a 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis (stage 0-III)
* Treated at Cleveland Clinic by medical oncologist, radiation oncologist, and/or breast surgeon Patients currently undergoing treatment or have completed active treatment (surgery, radiation or chemotherapy) within past 5 years.
* Able and willing to participate in art or music therapy programs at Maroone Cancer Center
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Ability to read and write in English
* Performance status 0 or 1 as per ECOG scale

Exclusion Criteria:

* No prior history of breast cancer
* History of metastatic disease (Stage IV)
* Not being followed by medical oncologist, radiation oncologist, and/or breast surgeon at Cleveland Clinic
* Unable or unwilling to participate in art or music therapy program at Maroone Cancer Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy: Breast Cancer (FACT-B) questionnaire scores | Baseline
  Quality of life (QOL) as measured by Functional Assessment of Cancer Therapy: Breast Cancer (FACT-B) questionnaire. This is a validated survey, completed by the patient, consisting of 37 items, each scored on a 0-4, Likert scale (0 = "Not at all"; 4= "Very much"). Subscales include: Physical Well-Being (PWB) (score range: 0-28), Social/Family Well-Being (SWB) (score range: 0-28), Emotional Well-Being (EWB) (score range: 0-24), Functional Well-being (FWB) (score range: 0-28), and the additional breast cancer concerns (BCS) (score range: 0-40) all with higher scores indicating better outcomes. Total scale scores range from 0 to 148 with higher scores indicating better outcomes.
FACT-B questionnaire scores | At 30-days
  QOL as measured by FACT-B questionnaire scores. This is a validated survey, completed by the patient, consisting of 37 questions, each scored on a 0-4, Likert scale (0 = "Not at all"; 4= "Very much"). Subscales include: PWB (score range: 0-28), SWB (score range: 0-28), EWB (score range: 0-24), FWB (score range: 0-28), and BCS (score range: 0-40) all with higher scores indicating better outcomes. Total scale scores range from 0 to 148 with higher scores indicating better outcomes.
FACT-B questionnaire scores | At 90-days
  QOL as measured by FACT-B questionnaire scores. This is a validated survey, completed by the patient, consisting of 37 questions, each scored on a 0-4, Likert scale (0 = "Not at all"; 4= "Very much"). Subscales include: PWB (score range: 0-28), SWB (score range: 0-28), EWB (score range: 0-24), FWB (score range: 0-28), and BCS (score range: 0-40) all with higher scores indicating better outcomes. Total scale scores range from 0 to 148 with higher scores indicating better outcomes.
FACT-B questionnaire scores | At 180-days
  QOL as measured by FACT-B questionnaire scores. This is a validated survey, completed by the patient, consisting of 37 questions, each scored on a 0-4, Likert scale (0 = "Not at all"; 4= "Very much"). Subscales include: PWB (score range: 0-28), SWB (score range: 0-28), EWB (score range: 0-24), FWB (score range: 0-28), and BCS (score range: 0-40) all with higher scores indicating better outcomes. Total scale scores range from 0 to 148 with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Cognition (FACT-Cog) questionnaire scores | Baseline
  Cognition as measured by FACT-Cog questionnaire scores. This questionnaire contains 37 items, divided into four subscales: 1) patients' perceived cognitive impairments (score range: 0-72), 2) perceived cognitive abilities (score range: 0-28), 3) Noticeability or comments from others (score range: 0-16), and 4) impact of cognitive changes on QOL (score range: 0-16).
  Higher scores indicate worse perceived cognitive deficit. FACT-Cog sub-scores are studied on their own and not included in a "total score", as advised by the scoring guidelines
FACT-Cog questionnaire scores | At 30-days
  Cognition as measured by FACT-Cog questionnaire scores. This questionnaire contains 37 items, divided into four subscales: 1) patients' perceived cognitive impairments (score range: 0-72), 2) perceived cognitive abilities (score range: 0-28), 3) Noticeability or comments from others (score range: 0-16), and 4) impact of cognitive changes on QOL (score range: 0-16).
  Higher scores indicate worse perceived cognitive deficit. FACT-Cog sub-scores are studied on their own and not included in a "total score", as advised by the scoring guidelines
FACT-Cog questionnaire scores | At 90-days
  Cognition as measured by FACT-Cog questionnaire scores. This questionnaire contains 37 items, divided into four subscales: 1) patients' perceived cognitive impairments (score range: 0-72), 2) perceived cognitive abilities (score range: 0-28), 3) Noticeability or comments from others (score range: 0-16), and 4) impact of cognitive changes on QOL (score range: 0-16).
  Higher scores indicate worse perceived cognitive deficit. FACT-Cog sub-scores are studied on their own and not included in a "total score", as advised by the scoring guidelines
FACT-Cog questionnaire scores | At 180-days
  Cognition as measured by FACT-Cog questionnaire scores. This questionnaire contains 37 items, divided into four subscales: 1) patients' perceived cognitive impairments (score range: 0-72), 2) perceived cognitive abilities (score range: 0-28), 3) Noticeability or comments from others (score range: 0-16), and 4) impact of cognitive changes on QOL (score range: 0-16).
  Higher scores indicate worse perceived cognitive deficit. FACT-Cog sub-scores are studied on their own and not included in a "total score", as advised by the scoring guidelines
Generalized Anxiety Disorder-7 item (GAD-7) scores | Baseline
  Self-reported anxiety as measured by GAD-7 scores. Scoring is scaled, as follows: 0 indicates "not at all", 1 indicates "several days", 2 indicates "more than half of the days", and 3 indicates "nearly every day for anxiety frequency".
Generalized Anxiety Disorder-7 item (GAD-7) scores | At 30-days
  Self-reported anxiety as measured by GAD-7 scores. Scoring is scaled, as follows: 0 indicates "not at all", 1 indicates "several days", 2 indicates "more than half of the days", and 3 indicates "nearly every day for anxiety frequency".
Generalized Anxiety Disorder-7 item (GAD-7) scores | At 90-days
  Self-reported anxiety as measured by GAD-7 scores. Scoring is scaled, as follows: 0 indicates "not at all", 1 indicates "several days", 2 indicates "more than half of the days", and 3 indicates "nearly every day for anxiety frequency".
Generalized Anxiety Disorder-7 item (GAD-7) scores | At 180-days
  Self-reported anxiety as measured by GAD-7 scores. Scoring is scaled, as follows: 0 indicates "not at all", 1 indicates "several days", 2 indicates "more than half of the days", and 3 indicates "nearly every day for anxiety frequency".
Patient Health Questionnaire-9 item (PHQ-9) scores | Baseline
  Self-reported depression as measured by PHQ-9 scores. A score of 0-4 indicates no depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, and a score of 15 or more indicates severe depression
Patient Health Questionnaire-9 item (PHQ-9) scores | At 30-days
  Self-reported depression as measured by PHQ-9 scores. A score of 0-4 indicates no depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, and a score of 15 or more indicates severe depression
Patient Health Questionnaire-9 item (PHQ-9) scores | At 90-days
  Self-reported depression as measured by PHQ-9 scores. A score of 0-4 indicates no depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, and a score of 15 or more indicates severe depression
Patient Health Questionnaire-9 item (PHQ-9) scores | At 180-days
  Self-reported depression as measured by PHQ-9 scores. A score of 0-4 indicates no depression, a score of 5-9 indicates mild depression, a score of 10-14 indicates moderate depression, and a score of 15 or more indicates severe depression
Attitudes towards art/music scores | Baseline
  Intervention efficacy as measured by attitudes towards art/music, assessed in 4, 10-point Likert questions with scores ranging from 0 to 40, and higher scores indicating better attitudes.
  Age, race/ethnicity, marital status, no. of children (if any), occupation, time since diagnosis, current chemotherapy regimen, time since therapy initiated / completed, and attitudes towards art and music will be collected as variables, to assess whether these factors are significant predictors of intervention efficacy.
Attitudes towards art/music scores | At 30-days
  Intervention efficacy as measured by attitudes towards art/music, assessed in 4, 10-point Likert questions with scores ranging from 0 to 40, and higher scores indicating better attitudes.
Attitudes towards art/music scores | At 90-days
  Intervention efficacy as measured by attitudes towards art/music, assessed in 4, 10-point Likert questions with scores ranging from 0 to 40, and higher scores indicating better attitudes.
Attitudes towards art/music scores | At 180-days
  Intervention efficacy as measured by attitudes towards art/music, assessed in 4, 10-point Likert questions with scores ranging from 0 to 40, and higher scores indicating better attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Florida Weston, Case Comprehensive Cancer Center, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share manuscripts, presentations, and abstracts